CLINICAL TRIAL: NCT00200174
Title: Combined Estrogen Blockade of the Breast With Exemestane and Raloxifene in Postmenopausal Women With a History of Breast Cancer Who Have No Clinical Evidence of Disease: A Pilot Chemoprevention Trial
Brief Title: Combined Estrogen Blockade of the Breast With Exemestane and Raloxifene in Postmenopausal Women With a History of Breast Cancer Who Have No Clinical Evidence of Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Pharmacia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 99-017; NCT00004247 (obsolete NCT alias)
Record Dates: First submitted 2005-09-09; First posted 2005-09-20 (Estimated); Last update posted 2023-07-05 (Actual); Status verified 2023-07

CONDITIONS: Breast Cancer
Keywords: Breast cancer; estrogen; postmenopausal
MeSH Terms: conditions — Breast Neoplasms

ARMS (2):
- A (Active Comparator): Raloxifene followed by combination therapy
  Interventions: Drug: Raloxifene followed by combination therapy
- B (Active Comparator): Exemestane followed by combination therapy
  Interventions: Drug: Exemestane followed by combination therapy

INTERVENTIONS:
Drug: Raloxifene followed by combination therapy — Patients will be randomized to either Raloxifene at 60mg P.O. (each day) for 2 weeks (time designated: week- 2) After two weeks of single agent therapy, patients will be started on combination therapy with oral raloxifene (60mg/day) and oral exemestane (25mg/day) (time designated week 0), and continued on both drugs for one year (month 12). Patients will be required to start supplemental calcium (900-1500 mg/day) plus vitamin D (400-600 units/day) P.O. each day during week 0.
  Arms: A
Drug: Exemestane followed by combination therapy — Patients will be randomized to Exemestane at 25mg P.O. for 2 weeks (time designated: week- 2) After two weeks of single agent therapy, patients will be started on combination therapy with oral raloxifene (60mg/day) and oral exemestane (25mg/day) (time designated week 0), and continued on both drugs for one year (month 12). Patients will be required to start supplemental calcium (900-1500 mg/day) plus vitamin D (400-600 units/day) P.O. each day during week 0.
  Arms: B

SUMMARY:
The purpose of this research study is to learn about the effects of two drugs when they are given together. The names of the drugs are raloxifene and exemestane.

Raloxifene is a drug that is related to estrogen. In the liver and bone, it acts like estrogen. In the breast and uterus it acts like an anti-estrogen. It has been used in postmenopausal women to prevent a disease called osteoporosis. This is a disease that decreases bone strength over many years and may finally lead to bone fractures. In a group of women who were taking the drug, it also seemed to decrease the chances of breast cancer and possibly endometrial cancer (cancer of the uterus). Therefore, we want to study it further to see if it prevents breast cancer. We also want to find out if it may be even better in preventing breast cancer if it is given with another drug.

The other drug in this trial is exemestane. Exemestane is a type of drug that works to decrease estrogen levels in postmenopausal women. This type of drug is used in women for the treatment of breast cancer. Before we can decide if the two drugs combined are better for preventing breast cancer, we must first test these drugs together to make sure that they are safe. This safety testing is the purpose of this trial.

DETAILED DESCRIPTION:
The objectives of this project are to investigate the safety and toxicity of the combination of raloxifene, a selective estrogen receptor modulator (SERM), with exemestane, a new steroidal aromatase inhibitor, in postmenopausal women with a history of breast cancer who have no clinical evidence of disease. The study cohort will consist of postmenopausal women with a history of AJCC Stage 0, I, II, or III breast cancer after completion of all planned adjuvant therapy. The study cohort is limited to patients who have not already received anti-estrogen therapy as part of post-operative adjuvant treatment. Patients with a history of invasive ER- and/or PR-positive breast cancer are eligible only if they have not received an anti-estrogen as part of adjuvant therapy, and they are at least 2 years from the time of their primary surgery.

Tamoxifen has been shown to reduce the incidence of contralateral breast cancer regardless of the estrogen expression of the primary tumor and may therefore be offered as a chemopreventive agent to patients who have not received an anti-estrogen in the adjuvant setting. This population of patients is also a reasonable cohort in which to test other chemoprevention regimens. Our hypothesis is that the combination of raloxifene and exemestane may offer an alternative treatment for chemoprevention that may prove to be more effective than an anti-estrogen alone.

Endpoints of the study are to determine whether the combination of raloxifene and exemestane is safe and tolerable with respect to:

1. markers of bone turnover and bone mineral density
2. the serum lipoprotein profile
3. quality of life (in particular, symptoms of estrogen deficiency)
4. pharmacokinetics and pharmacodynamics of both drugs.

We will also determine the feasibility of using mammography and breast MRI imaging to assess the effects of the combination on radiographic breast density.

As part of a correlative laboratory study of breast biopsy material, women may undergo an optional biopsy of their unaffected breast. Breast biopsy material will be evaluated both pre- and 3 months post-treatment to determine whether the combination will have an impact on breast tissue aromatase activity and breast tissue estrogen levels, and potential surrogate endpoint biological markers.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women with a history of AJCC Stage 0, I, II or III breast cancer, with no clinical evidence of disease, after completion of all planned adjuvant therapy. Patients must not have received anti-estrogen therapy as part of their adjuvant treatment. Patients with a history of invasive ER- and/or PR-positive breast cancer are eligible only if they have not received an anti-estrogen as part of adjuvant therapy, and they are at least 2 years from the time of their primary surgery.
* Patients must have completed all planned adjuvant therapy, including surgery, chemotherapy, and radiation therapy, at least 4 weeks prior to treatment. There is no limit as to the amount of time that may have passed since completion of adjuvant therapy and initiation of treatment.
* Patients must be postmenopausal, as defined by either:

  1. No spontaneous menses for at least 5 years; women who have had a hysterectomy in this group, but have intact ovaries must have luteinizing hormone (LH) and follicle-stimulating hormone (FSH) levels within the postmenopausal range
  2. Spontaneous menses within the past 5 years, but amenorrheic (e.g. spontaneous or secondary to chemotherapy, radiation therapy or hysterectomy) for at least 12 months, and luteinizing hormone (LH) and follicle-stimulating hormone (FSH) levels within the postmenopausal range
  3. Bilateral oophorectomy
* Patients must have a history of breast cancer confirmed by the Department of Pathology at Memorial Sloan-Kettering Cancer Center.
* Patients must be at least 18 years old, and must be able to give written informed consent.
* Karnofsky performance status > 80%.
* Laboratory parameters:

WBC =>3.0 x 106 cells/ml serum bilirubin <= 1.5 mg/dl serum creatinine <= 1.5 mg/dl serum AST (SGOT) <= 2x upper institutional normal CEA and CA15-3 within institutional normal limits

Exclusion Criteria:

* Prior history of bilateral mastectomy.
* Prior history of ovarian or endometrial cancer.
* Prior or current history of osteoporosis, as defined by a lumbar-spine bone mineral density < 2.5 SD below the mean value for normal premenopausal women.
* Use of bisphosphonates or calcitonin within the past 3 months.
* Prior history of venous thrombosis or pulmonary embolism.
* Patients with unstable angina or New York Heart Association Class III or IV heart disease.
* Prior hormonal therapy within the past 3 months.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 1999-07; Primary Completion 2003-07 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the clinical safety and toxicity of raloxifene in combination with exemestane in postmenopausal women with a hx of AJCC Stage 0, I, II, or III breast cancer, who have no clinical evidence of disease, after completion of all planned adjuvant | 1 year

SECONDARY OUTCOMES:
To determine the feasibility of using mammography and breast MRI imaging to assess the effects of raloxifene plus exemestane on radiographic breast density. | baseline and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Maura Dickler, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://mskcc.org